CLINICAL TRIAL: NCT04649528
Title: Digitally Assisted High-intensity Interval Training in Inflammatory Rheumatic Disease Patients: Treatment by Man or Machine?
Brief Title: HIIT for Inflammatory Rheumatic Disease: Man vs Machine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHRevma1
Record Dates: First submitted 2020-11-19; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Inflammatory Rheumatism
Keywords: VO2max; Cardiovascular health; Quality of life; Endurance exercise
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Intervention Model Description: Randomized trial
Who Masked: Investigator
Masking Description: The exercise physiologist performing the maximal oxygen uptake pre and posttests was blinded with reguards to which intervention group the participants had been assigned.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised HIIT (Experimental): Exercise intervention, 20 supervised by healthcare professional
  Interventions: Behavioral: Effective endurance 4x4 training - Supervised
- APP HIIT (Experimental): Exercise intervention, 20 self-monitored assisted by a mobilephone application
  Interventions: Device: Effective endurance 4x4 training - APP

INTERVENTIONS:
Behavioral: Effective endurance 4x4 training - Supervised — Exercise intervention utilizing 4x4min aerobic high-intensity interval training
  Arms: Supervised HIIT
Device: Effective endurance 4x4 training - APP — Exercise intervention utilizing 4x4min aerobic high-intensity interval training
  Arms: APP HIIT

SUMMARY:
The purpose of this study is to compare two modes of delivering high-intensity interval training (HIIT) in a population with inflammatory rheumatic disease over 10 weeks. One group will recieved HIIT supervised by a healthcare professional, the other group will perform self-monitored HITT with guidance by a smarthpone application.

DETAILED DESCRIPTION:
People with inflammatory rheumatic diseases (IRS) such as rheumatoid arthritis (RA), spondyloarthritis (SpA) and systemic lupus erythematosus (SLE) have been shown to have reduced cardiovascular fitness and quality of life than the general population. Cardiovascular health is the single most important factor of total mortality. It has been shown previously that individuals with IRS tolerate both endurance training, resulting in improvement in function and cardiovascular health while also having a positive effect on disease activity measured through inflammation, pain, joint health and fatigue. In recent years, studies have also been conducted that demonstrate both the safety and effect of aerobic 4x4min high-intensity interval training (HIIT) for patients with IRS.

This study will involve an intervention period consisting of 20 HIIT sessions. Participants are randomized into one of two training groups. One group will perform HIIT under the supervision of a healthcare professional. The other group will perform the same HIIT training with identical instructions, however they will be self-monitored with the aid and guidance of a mobilephone application.

The purpose of the intervention is to increase maximum oxygen uptake and improve quality of life. The intervention period will consist of 2 weekly sessions lasting approximately 35 minutes performed on non-consecutive days. The endurance training will consist of 4 intervals of 4 minutes duration, separated by a 3-4 minute active break and follows the principle of intensive aerobic interval training. Before and after the training period, identical testing (approximately 30-40 min) will be performed by both intervention groups. The testing will include measurements of work economy and maximal oxygen uptake in an endurance test. Additionally, quality of life questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

- Inflammatory rheumatic disease

Exclusion Criteria:

* Inability to complete the testing procedures
* Pregancy
* Not able to perform exercise intervention
* Planed surgeries or other plans during initial exercise intervention period than directly will effect the testing or training.
* Access to a smartphone
* Less than 80% compliance of planned training sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Change in physiological measures | At baseline and after 10 weeks of HIIT
  Maximal oxygen uptake

SECONDARY OUTCOMES:
Change in health-related quality of life | At baseline and after 10 weeks of HIIT
  Questionnaire (Norwegian RAND-36), scoring on a 0-100 scale with higher scores identifying better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Helgerud, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Myworkout - Medical Rehabilitation Clinic, Trondheim, Please Select, Norway

REFERENCES:
- [Derived] Haglo H, Wang E, Berg OK, Hoff J, Helgerud J. Smartphone-Assisted High-Intensity Interval Training in Inflammatory Rheumatic Disease Patients: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Oct 21;9(10):e28124. doi: 10.2196/28124. PMID 34673536